CLINICAL TRIAL: NCT00281944
Title: A Multi-Center Phase Ib Study of Oxaliplatin (NSC #266046) in Combination With Fluorouracil and Leucovorin in Pediatric Patients With Advanced Solid Tumors
Brief Title: Combination Chemotherapy in Treating Young Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01051; 04-0336; MSKCC-040336; CDR0000454709; NCI-6952; POETIC-COMIRB-040336
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Childhood Central Nervous System Choriocarcinoma; Childhood Central Nervous System Embryonal Tumor; Childhood Central Nervous System Germ Cell Tumor; Childhood Central Nervous System Germinoma; Childhood Central Nervous System Mixed Germ Cell Tumor; Childhood Central Nervous System Teratoma; Childhood Central Nervous System Yolk Sac Tumor; Recurrent Childhood Brain Stem Glioma; Recurrent Childhood Central Nervous System Embryonal Tumor; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: interventions — Oxaliplatin; Fluorouracil; Leucovorin; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

ARMS (1):
- Treatment (oxaliplatin, leucovorin calcium, fluorouracil) (Experimental): Patients receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 followed by fluorouracil IV continuously over 46 hours on days 1-2. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: oxaliplatin; Drug: fluorouracil; Drug: leucovorin calcium; Other: pharmacological study; Procedure: positron emission tomography; Procedure: computed tomography

INTERVENTIONS:
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Procedure: positron emission tomography — Undergo PET scan
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Procedure: computed tomography — Undergo PET/CT scan
  Other Names: tomography, computed

SUMMARY:
This phase I trial is studying the side effects and best dose of oxaliplatin when given together with leucovorin and fluorouracil in treating young patients with advanced solid tumors. Drugs used in chemotherapy, such as oxaliplatin, leucovorin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the dose-limiting toxicities (DLT) and maximum tolerated dose (MTD) of oxaliplatin when given together with fluorouracil and leucovorin calcium in pediatric patients with recurrent or refractory solid tumors, including tumors of the CNS.

SECONDARY OBJECTIVES:

I. Determine the pharmacokinetic properties of oxaliplatin in this pediatric patient population.

II. Correlate alterations in accumulation of fludeoxyglucose F 18 with tumor response in those patients who can readily undergo a positron emission tomography (PET) or PET/CT scan.

III. Assess the safety profile of this regimen in these patients. IV. Evaluate any preliminary evidence of anti-tumor activity of this regimen in these patients.

OUTLINE: This is an open-label, multicenter, dose-escalation study of oxaliplatin. Patients are stratified according to solid tumor type (non-CNS vs CNS).

Patients receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 followed by fluorouracil IV continuously over 46 hours on days 1-2. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of oxaliplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed malignant solid tumor, including tumors of the CNS, that has progressed despite standard therapy or for which no effective standard therapy is known

  * Patients with brainstem glioma or intrinsic pontine glioma do not need biopsy proof of the diagnosis if imaging studies are consistent with the diagnosis
* Measurable or nonmeasurable disease
* No pleural effusion or ascites causing respiratory compromise (≥ grade 2 dyspnea)
* ECOG performance status (PS) 0-2 for patients ≥ 16 years of age
* Karnofsky PS ≥ 40% for patients > 10 years of age
* Lansky Play Scale ≥ 40% for patients ≤ 10 years of age
* Peripheral absolute neutrophil count (ANC) ≥ 1,000/mm^3
* Platelet count ≥ 75,000/mm^3 (transfusion independent)
* Hemoglobin ≥ 8.5 g/dL (transfusion permitted)
* Serum creatinine ≤ 1.5 times upper limit of normal (ULN)
* Creatinine clearance OR radioisotope glomerular filtration rate > 60mL/min
* Total bilirubin < 1.5 mg/dL
* ALT and AST ≤ 2.5 times ULN (5 times ULN if liver involvement with primary tumor)
* Ejection fraction ≥ 50% OR shortening fraction ≥ 28%
* Life expectancy of > 8 weeks
* No radiological evidence of pulmonary fibrosis, interstitial pneumonia, or extensive and symptomatic interstitial fibrosis of the lung

  * Room air oxygen saturation ≥ 90% at altitudes ≥ 5,000 feet OR ≥ 93% at altitudes < 5,000 feet
  * DLCO > 50% of predicted (for patients who received prior bleomycin and are able to comply with pulmonary function testing)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to platinum or oxaliplatin as well as other agents used in study treatment
* No other serious or poorly controlled social circumstance, psychiatric illness, or medical condition including, but not limited to, the following: ongoing or active infection, uncontrolled seizure disorder, uncontrolled symptomatic congestive heart failure, or cardiac arrhythmia that could be exacerbated by or complicate compliance with study therapy
* No HIV-positive patients
* Recovered from prior therapy

  * No persistent toxicities from previous therapies ≥ grade 2

    * Stable grade 3 neurotoxicity is allowed in patients with CNS tumors only who have a baseline neurotoxicity due to primary tumor involvement or postoperative complications
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* At least 4 weeks since prior local radiotherapy (small port)
* At least 6 months since prior craniospinal irradiation, irradiation to ≥ 50% of the pelvis, or other substantial bone marrow irradiation, including total body irradiation
* No previous treatment with oxaliplatin
* At least 14 days since prior biological therapy (including monoclonalantibody therapy)
* At least 7 days since prior retinoids, sargramostim (GM-CSF), or filgrastim (G-CSF)
* At least 14 days since prior pegfilgrastim
* No concurrent pegfilgrastim or GM-CSF
* Patients requiring steroids should be on stable or decreasing dose for ≥ 7 days prior to study entry, and must not be on more than 4 mg of dexamethasone (or equivalent) per day
* At least 4 weeks since prior major surgical procedure

  * Simple surgical procedures, including biopsy or central line placement or similar procedure, are allowed within 4 weeks of study entry if the patient has recovered to baseline
* At least 3 months since prior autologous or allogeneic stem cell transplantation

  * No concurrent immunosuppressive therapy
  * No evidence of ongoing graft versus host disease (GVHD)
* No concurrent use of other investigational agents
* No other concurrent anticancer therapies or agents
* No other concurrent chemotherapy, radiation therapy, or herbal medications or supplements

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2005-09; Primary Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
MTD based on the incidence of DLT as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v.) 3.0 | 14 days
DLT defined as any grade 3 or greater non-hematologic toxicity attributed to the combination of drugs in this regimen, despite maximal supportive care as assessed by NCI CTCAE v. 3 | 14 days

SECONDARY OUTCOMES:
Safety profile as assessed by NCI CTCAE v. 3.0 | 14 days
  Any incidence of adverse events will be recorded and classified according to body region and severity.
Tumor response based on PET or PET/CT scan | From baseline to 6 weeks
  Wilcoxon rank sum statistic will be used to assess whether tumor response is associated with the change in the PET SUV value.

CONTACTS AND LOCATIONS:
Overall Officials: Lia Gore, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States